CLINICAL TRIAL: NCT01415037
Title: High-frequency-ultrasound Annular Arrays for Ophthalmic Imaging
Brief Title: Annular Array Ultrasound in Ophthalmology
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Riverside Research Institute (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ronald H. Silverman, Professor of Ophthamlic Science, Columbia University
Other Study IDs: AAAF3057; R21EY024434 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-08-11 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Posterior Vitreous Detachment; Diabetic Retinopathy
Keywords: Annular Array Ultrasound; Ultrasound Exam; Posterior Vitreous Detachment; PVD; Diabetic Retinopathy
MeSH Terms: conditions — Vitreous Detachment; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Annular Array Ultrasound: Subject with possible or with known posterior vitreous detachment. Subjects with diabetic retinopathy will receive annular array ultrasound exam.
  Interventions: Procedure: annular array ultrasound exam

INTERVENTIONS:
Procedure: annular array ultrasound exam — For this research study you will be asked to sit in a chair. You will be given 2 drops of a numbing solution. The ultrasound camera will be enclosed in a sterile membrane and will be placed gently upon your eye. You may be asked to gaze at a light source while measurements are being made. The procedure will last about 10-15 minutes from start to finish.

SUMMARY:
The objective of this research is to improve the care of ocular disease and disorders, in particular the changes in the eye associated with diabetes, by providing clinicians with dramatically improved ultrasonic images of the entire eye. The research combines advanced high-frequency, high-resolution ultrasonic annular arrays transducers with new processing techniques designed to overcome several limits that have been reached with conventional high frequency ultrasound systems. The investigators propose that diagnosis of eye diseases using annular arrays can be more effective than the conventional ultrasound images by at least 50%; i.e., that for every 2 posterior vitreous detachments detected conventionally, 3 will be detected with the annular arrays.

DETAILED DESCRIPTION:
The goal of this study is to develop and evaluate advanced annular-array transducer technology for rapid, high-definition imaging. The study will assess high frequency ultrasound (HFU, 40 & 20 MegaHertz) annular arrays in imaging posterior vitreous detachments (PVDs) associated with diabetic retinopathy, the leading cause of blindness in the US working-age population according to Prevent Blindness America. Current HFU instruments do not use linear arrays for such applications because of a variety of technical and cost reasons. Instead, current HFU instruments use mechanically scanned, single-element transducers, which provide fine-resolution images over a very limited depth of field (DOF). For ophthalmic applications, a shallow DOF causes most ocular anatomy to be imaged with poor definition compared to the in-focus region; therefore, because only a small portion of the eye is in focus at a given time, detection and assessment of ocular conditions such as PVD are prone to inaccuracies and false-negative determinations. Annular-array transducers offer a promising approach to significantly extend DOF and to increase the depth range over which fine-lateral resolution is provided. The investigators will validate system performance using animal experiments and human-subject examinations. First, in vivo animal experiments will be conducted to evaluate a 40-MegaHertz (MHz) annular array for anterior-segment imaging and a 20-MHz annular array for posterior segment and full-globe imaging. The investigators will test the hypothesis that 20-MHz annular arrays improve detection of PVD. Validation of this hypothesis will significantly improve our ability to assess disease status in diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* over age 60
* people with diabetic retinopathy or posterior vitreous detachments

Exclusion Criteria:

* under age 60

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University-based Ophthalmology Practice
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in detection of posterior vitreous detachment: 20MHz annular array versus 10MHz single element | Subjects will be examined with both the 20MHz annular array and 10MHz single element ultrasound during the same exam, approximately 30 minutes in duration.
  The investigators will examine eyes with both conventional 10MHz ultrasound and a 20MHz annular array with synthetic focusing. The investigators will evaluate and compare images acquired with both techniques and determine their relative efficacy in visualizing the presence or absence of posterior vitreous detachment.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Silverman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Mamou J, Aristizabal O, Silverman RH, Ketterling JA, Turnbull DH. High-frequency chirp ultrasound imaging with an annular array for ophthalmologic and small-animal imaging. Ultrasound Med Biol. 2009 Jul;35(7):1198-208. doi: 10.1016/j.ultrasmedbio.2008.12.017. Epub 2009 Apr 25. PMID 19394754
- [Background] Mamou J, Ketterling JA, Silverman RH. Chirp-coded excitation imaging with a high-frequency ultrasound annular array. IEEE Trans Ultrason Ferroelectr Freq Control. 2008 Feb;55(2):508-13. doi: 10.1109/TUFFC.2008.670. PMID 18334358
- [Background] Silverman RH, Ketterling JA, Coleman DJ. High-frequency ultrasonic imaging of the anterior segment using an annular array transducer. Ophthalmology. 2007 Apr;114(4):816-22. doi: 10.1016/j.ophtha.2006.07.050. Epub 2006 Nov 30. PMID 17141314
- [Background] Filoux E, Sampathkumar A, Chitnis PV, Aristizabal O, Ketterling JA. High-frequency annular array with coaxial illumination for dual-modality ultrasonic and photoacoustic imaging. Rev Sci Instrum. 2013 May;84(5):053705. doi: 10.1063/1.4804636. PMID 23742556
- [Background] Lethiecq M, Lou-Moeller R, Ketterling J, Levassort F, Tran-Huu-Hue LP, Filoux E, Silverman RH, Wolny WW. Non-planar pad-printed thick-film focused high-frequency ultrasonic transducers for imaging and therapeutic applications. IEEE Trans Ultrason Ferroelectr Freq Control. 2012 Sep;59(9):1976-82. doi: 10.1109/TUFFC.2012.2416. PMID 23007770
- [Result] Mamou J, Wa CA, Yee KM, Silverman RH, Ketterling JA, Sadun AA, Sebag J. Ultrasound-based quantification of vitreous floaters correlates with contrast sensitivity and quality of life. Invest Ophthalmol Vis Sci. 2015 Jan 22;56(3):1611-7. doi: 10.1167/iovs.14-15414. PMID 25613948
- [Result] Silverman RH, Ketterling JA, Mamou J, Lloyd HO, Filoux E, Coleman DJ. Pulse-encoded ultrasound imaging of the vitreous with an annular array. Ophthalmic Surg Lasers Imaging. 2012 Jan-Feb;43(1):82-6. doi: 10.3928/15428877-20110901-03. Epub 2011 Sep 8. PMID 21902166